CLINICAL TRIAL: NCT03440762
Title: Evaluation of a Community-Placed Atrial Fibrillation Screening and Education Program
Brief Title: Atrial Fibrillation Screening and Education Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Heart Rhythm Society (Unknown)
Responsible Party: Principal Investigator, Pamela J. McCabe, R.N., Ph.D., Nurse Scientist, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 17-005031
Record Dates: First submitted 2018-02-01; First posted 2018-02-22 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation
Keywords: Screening; Education; AFib Awareness; Stroke prevention
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Single group pre-post educational intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AF awareness education (Other): AF awareness education face to face
  Interventions: Behavioral: AF awareness education

INTERVENTIONS:
Behavioral: AF awareness education — Participants will receive education about a description of AF, complications, recognition of signs and symptoms of AF, pulse taking, and how to recognize an irregular pulse

SUMMARY:
The purpose of this study is to evaluate the outcomes of a community placed atrial fibrillation (AF) screening and education program

DETAILED DESCRIPTION:
Background/significance: Atrial fibrillation (AF) is a global epidemic that accounts for 15%-20% of 795,000 strokes occurring annually in the US, at a cost of $3.2 billion per year. Atrial fibrillation-related stroke will rise with the aging population and places enormous strain on healthcare resources and quality of life; yet they are highly preventable, by early detection of AF. Timely treatment reduces AF-related stroke risk by 68%, yet treatment is often delayed because people may not recognize the symptoms of AF or may be asymptomatic. Given the number of people at risk for development of AF and the dire consequences of untreated AF, efforts to promote early detection of AF through proactive screening of older adults at risk for AF have been successfully undertaken in Europe and Australia. However, little is known about the outcomes of conducting programs to screen for and educate people about AF in community settings in the US.

Purpose: The purpose of this descriptive pragmatic study to evaluate the outcomes of a community placed AF screening and education program. Primary outcomes include feasibility, number of participants who screen positive for AF, and changes in participants' Knowledge, Attitudes, and Beliefs about Atrial Fibrillation Self-Monitoring (KABAF-SM) scores from baseline to two-weeks after enrollment.

Methods: Up to 250-participants who have at least two risk factors for developing AF and have no previous diagnosis of AF will be recruited from Midwest community settings and will be screened for AF using a mobile ECG recorder and will receive written information sheet about AF. A portion (up to 125) of those 250 participants will be invited to complete the KABAF-SM at baseline and 2-weeks after enrollment. Participants will have the option to participate in a variety of AF educational activities to reinforce and enhance the written information. Participants will be surveyed about their perceptions of the educational program after the screening and participating in the educational activities.

Evaluation methods: Descriptive statistics will be used to analyze feasibility (enrollment numbers, participants perception of the value of the educational activities, time required for study procedures,and AF detection.T-tests will be used to test for differences between KABAF-SM baseline and two-week scores for those who completed the KABAF-SM.

ELIGIBILITY:
Inclusion :

Any two of the following:

* Hypertension
* Diabetes
* Sleep apnea
* Obesity
* Age > 75 years
* Peripheral arterial disease
* Female

Exclusion :

* Previous diagnosis of atrial fibrillation or atrial flutter
* Uncompensated visual impairment
* Uncompensated hearing impairment
* Inability to communicate verbally in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Feasibility-number enrolled | 5 months
  number of participants enrolled
Feasibility-time required for study procedure | 5 months
  Number of minutes require to perform mobile ECG
Participants' perception of the usefulness of the Learning Station activities | 5 months
  The outcome will be measured by the Participant Perception of Learning Station Activities survey. This survey is an investigator developed 9-item Survey that asks participants to rate how useful learning activities were to increase their knowledge about atrial fibrillation and to what extent their knowledge about atrial fibrillation has increased after participating in the Learning Station activities. Psychometric testing has not been performed on this survey.

SECONDARY OUTCOMES:
Change in knowledge attitude, and beliefs scores about AF self monitoring from baseline | 5 months
  Knowledge, attitudes, beliefs about self-monitoring for AF signs and symptoms will be measured by the Knowledge Attitudes and Beliefs about Atrial Fibrillation Self-Monitoring (KABAF-SM) instrument.The KABAF-SM is a 40-item instrument that measures knowledge of AF symptoms (8 items yes/no response, score range 0-8); symptoms not related to AF (6 items yes/no response, score range 0-6); and Likert- responses items (strongly disagree-1 to strongly agree-4) for beliefs about the participant's risk for developing AF(5 items), seriousness of AF,(4 items) benefits (5 items), and barriers (5 items) to monitoring for signs and symptoms of AF. Total score range for the Likert items is 14-56. Perceived confidence is measured by 7 items, rated from 0-10 (score range, 0-70) for ability to self-monitor for signs and symptoms of AF. Higher scores reflect more knowledge and more accurate beliefs and positive attitudes toward self-monitoring.
Number of cases of atrial fibrillation detected with portable ECG | 5 months
  The Alive Cor portable ECG recorder will be used to detect atrial fibrillation. The device displays the participants rhythm as normal sinus, possible or probable atrial fibrillation, or unable to analyze

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J McCabe, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials